CLINICAL TRIAL: NCT03873935
Title: Evaluation of Vitamin D on Periodontal and Cardiovascular Diseases Progression
Brief Title: Vitamin D in Periodontal and Cardiovascular Disease Progression
Status: Completed | Type: Observational
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Gaetano Isola, DDS, PhD, Principal Investigator, University of Messina
Other Study IDs: #17-09
Record Dates: First submitted 2019-03-09; First posted 2019-03-14 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control: Healthy subjects
  Interventions: Other: Evaluation of periodontal status
- Periodontitis: Patients with periodontal disease
  Interventions: Other: Evaluation of periodontal status
- Cardiovascular: Patients with cardiovascular disease
  Interventions: Other: Evaluation of periodontal status
- Periodontitis+Cardiovascular: People with both cardiovascular and periodontitis
  Interventions: Other: Evaluation of periodontal status

INTERVENTIONS:
Other: Evaluation of periodontal status — Clinical examination

SUMMARY:
Vitamin D has been considered to possess anti-inflammatory and antimicrobial activity which may be a link for the known interaction of periodontitis (CP) and coronary heart disease (CHD). This study investigated the association between serum vitamin D levels and periodontitis in patients with CP and with CHD. Furthermore, the objective was to determine if periodontitis and CHD had an impact on serum vitamin D levels.

DETAILED DESCRIPTION:
Using a cross-sectional design, a total of 39 patients with CP, 38 patients with CHD, 38 patients with both CP and CHD, and 37 healthy subjects will enrolled in the present study.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least twenty teeth
* CP with a minimum of 40% of sites with a clinical attachment level (CAL) ≥2mm and probing depth (PD) ≥4mm;
* Presence of at least ≥2 mm of crestal alveolar bone loss verified on digital periapical radiographs
* Presence of ≥40% sites with bleeding on probing (BOP)

Exclusion Criteria:

* Intake of contraceptives
* Intake of immunosuppressive or anti-inflammatory drugs throughout the last three months prior to the study
* Status of pregnancy or lactation
* Previous history of excessive drinking
* Allergy to local anaesthetic
* Intake of drugs that may potentially determine gingival hyperplasia such as Hydantoin, Nifedipine, Cyclosporin A or similar drugs.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thus, for this study, at least of 39 patients with CP, 38 patients with CHD, 38 patients with both CP and CHD, and 37 healthy subjects will finally enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment level | 1 year
  Clinical Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — University of Messina
Locations (1):
- University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 1 year
Access Criteria: Pubmed website